CLINICAL TRIAL: NCT05897944
Title: Creating and Assessing a Voice Dataset for Automated Classification of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Excellence Center at Linköping - Lund in Information Technology (ELLIIT) (Unknown)
Responsible Party: Principal Investigator, Johan Sanmartin Berglund, Professor, MD, PhD, Blekinge Institute of Technology
Other Study IDs: BTH-6.1.1-0074-2023
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Automatic; Classification; COPD; Machine Learning; Mobile phone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Participants with clinically diagnosed Chronic obstructive pulmonary disease. Total 34 recruitment, 18 Female, 16 Male
  Interventions: Other: COPD
- HC: Participants without Chronic obstructive pulmonary disease diagnosis. Total 38 recruitment, 20 Female, 18 Male
  Interventions: Other: COPD

INTERVENTIONS:
Other: COPD — A data set consisting of information from COPD and HC groups will be used to experiment with the classification performance of several Machine Learning techniques.
  Other Names: HC

SUMMARY:
This work aims to evaluate whether voice recordings collected from patients diagnosed with COPD and healthy control groups can be used to detect the disease using machine learning techniques.

DETAILED DESCRIPTION:
Voice data and sociodemographic data on gender and age will be collected through the "VoiceDiganostic" application from the company Voice Diagnostic, which allows one to participate without location dependency. Participants with a diagnosis will be marked as the COPD group, and others will be marked as the healthy control group. Private information such as known comorbidities, personal security numbers, health parameters and communication information will be separately noticed in a participation table for each group.

The collected data will be transformed into mathematical vocal measures called voice features. A dataset consisting of voice features in conjunction with demographics and health data will be constructed for further usage as an input to ML techniques.

Descriptive statistical analysis will be held on attributes containing information on input data and gained outcomes from ML algorithms. The achieved results will be presented in the form of summary tables and graphs.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old and older.

Exclusion Criteria:

* being under 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data will be collected from participants 18 years old and older with and without COPD diagnosis will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | Week 51
  Binary detection performance of the ML algorithm
Input data importance scale | Week 51
  Features used as input data will be ranked from most important to less important one.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sanmartin Berglund, MD, PhD, Principal Investigator — Blekinge Institute of Technology
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Blekinge County, Sweden

IPD SHARING:
Plan to Share IPD: No
Participant data can not be shared due to the GDPR. However, the dataset created can be available upon request from the institution.

REFERENCES:
- [Derived] Idrisoglu A, Dallora AL, Cheddad A, Anderberg P, Jakobsson A, Sanmartin Berglund J. COPDVD: Automated classification of chronic obstructive pulmonary disease on a new collected and evaluated voice dataset. Artif Intell Med. 2024 Oct;156:102953. doi: 10.1016/j.artmed.2024.102953. Epub 2024 Aug 15. PMID 39222579